CLINICAL TRIAL: NCT06385028
Title: Personalized Physical Activity Promotion in Osteoarthritis Patients Using a Smartphone-based Solution
Brief Title: Physical Activity Promotion in Osteoarthritis Patients
Acronym: PIANISSIMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Œuvre Nationale de Secours Grande Duchesse Charlotte (Unknown)
Responsible Party: Principal Investigator, Laurent Malisoux, PhD, Group leader, Luxembourg Institute of Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20230213_PIANISSIMO
Record Dates: First submitted 2024-04-23; First posted 2024-04-25 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis
Keywords: physical activity promotion; daily steps; connected devices; knee; hip
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Pilot feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical activity promotion (Experimental): The entire population will receive the physical activity promotion intervention, composed of weekly goal setting and daily notification with information about physical activity and sedentary behavior.
  Interventions: Behavioral: Physical activity promotion

INTERVENTIONS:
Behavioral: Physical activity promotion — The intervention will be delivered through a phone application: each week, the participant will define a new daily step goal for the following week. Then he/she will receive daily notifications (except Sundays) about physical activity, sedentary behavior and their consequences on general health and osteoarthritis specifically. These notifications are designed to promote physical activity in this specific population.

SUMMARY:
The main purpose of this project is to promote physical activity in patients with osteoarthritis. More specifically, this study aims to test the acceptability of an app to promote physical activity in the target population, and consequently the feasibility of such an approach.

A mobile phone application - namely PIANISSIMO - will be developed specifically for this project. It aims to spread knowledge on the benefits of physical activity and collect data on how this knowledge can induce behavior changes toward a more physically active lifestyle.

The intervention is delivered via the app, which will send daily notifications on physical activity and sedentary behavior, and ask the participants to set their weekly goal (i.e., daily steps). The app will also collect daily steps count and ask the participant to fill in questionnaire on pain once a week.

DETAILED DESCRIPTION:
Osteoarthritis patients will be recruited from the general population living or working in Luxembourg.

The PIANISSIMO study is a feasibility pilot study. Thus, it is a single-group study, with the participants being their own controls. 150 participants with osteoarthritis will be included. For this study, a mobile application will be developed. It will include self-administered questionnaires, allow physical activity data collection, and deliver the intervention (goal setting, data feedback, notifications to the user and self-completion questionnaires). The intervention will last 6 months, with a further 6-month follow-up.

After signing the explicit consent and data protection notice, participants will encode data and information about individual and chronic pain characteristics, sport history, general health status: Individual questionnaire will include demographic data and general health status. The osteoarthritis pain questionnaire focuses on disease history and evaluation that will include a SF-WOMAC questionnaire. In order to deliver the same intervention for every participant, sham notifications will be send the first week, until the next Sunday for the first goals to be set. First real notification will be send the first Monday after the registration to the study.

The daily step count will be collected in background during the whole study. Then the intervention will be delivered though the phone application: each week, the participant will define a new daily step goal for the following week. Then he/she will receive daily notifications (except Sundays) about physical activity, sedentary behaviour and their consequences on general health and osteoarthritis specifically.

He/she will also be asked to fill in a pain questionnaire once a week. The participant can also spontaneously notify pain at any moment in the same questionnaire. At the end of each month, the participant will be asked about her/his functional status with the WOMAC-SF questionnaire.

At the end of the 6-month intervention, a questionnaire will be sent to the participant to evaluate the application.

During the 6-month follow-up, daily step count will still be collected in background, and pain questionnaires will be sent twice a month, but without any intervention delivered.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis patients, living or working in Luxembourg
* Signed informed consent form
* Adequate understanding of one of the study languages (English, French, or German)
* Stated willingness to comply with the study procedure consisting in completing the surveys and the digital physical activity intervention

Exclusion Criteria:

* Rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Weekly number of connections to the application over time | 0 to 6 months
  Adherence to the intervention will first be evaluated by the number of connections to the application for any reason.
Response rate to the weekly questionnaires over time | 0 to 6 months
  Adherence to the intervention will also be evaluated by the the response rate to the questionnaires (pain questionnaires and goal settings).

SECONDARY OUTCOMES:
Evolution of physical activity metrics | 0 to 6 months
  evolution of steps/day in response to the physical activity promotion intervention
influence of pain on physical activity practice | 0 to 6 months
  evolution of daily steps over the week following the pain report
influence of physical activity on pain report | 0 to 6 months
  record of daily steps over the week before the pain report

OTHER OUTCOMES:
long-term evolution of daily steps | 7 to 12 months
  evolution of steps/day after the end of the physical activity promotion intervention

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Malisoux, PhD, Principal Investigator — Luxembourg Institute of Health
Locations (1):
- Luxembourg Institute of Health, Strassen, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mura M, Portugal B, Mouton C, Grimm B, Seil R, Malisoux L. An app-based physical activity intervention for people with hip and knee osteoarthritis: protocol for the PIANISSIMO feasibility study. Pilot Feasibility Stud. 2025 Dec 5;12(1):5. doi: 10.1186/s40814-025-01744-z. PMID 41351123
- See also: Project page — https://www.lih.lu/en/research-scope/research-department/department-of-precision-health/physical-activity-sport-and-health/pianissimo/
- See also: Group page — https://www.lih.lu/en/research-scope/research-department/department-of-precision-health/physical-activity-sport-and-health/